CLINICAL TRIAL: NCT00484029
Title: A Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Nasal CO2 in the Symptomatic Treatment of Temporomandibular Disorders
Brief Title: Nasal Carbon Dioxide (CO2)for the Treatment of Temporomandibular Disorders (TMD)Related Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capnia, Inc. (Industry)
Responsible Party: Kristen Yen- Associate Director, Clinical, Capnia, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C301
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Temporomandibular Disorders; Pain; Headaches
Keywords: Temporomandibular Disorders; TMD; TMJ/TMD; Pain Management; Pain; Headaches
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain; Headache; Agnosia | interventions — Air

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nasal Carbon Dioxide
  Interventions: Drug: Nasal Carbon Dioxide
- 2 (Placebo Comparator): Air
  Interventions: Other: Air

INTERVENTIONS:
Drug: Nasal Carbon Dioxide — Nasal Carbon Dioxide
  Arms: 1
Other: Air — Air (Medical Grade)
  Arms: 2

SUMMARY:
This purpose of this study is to evaluate the safety and efficacy of treatment with nasal CO2 in the treatment of pain and other symptoms related to temporomandibular disorder (TMD).

DETAILED DESCRIPTION:
This is a randomized, controlled trial evaluating the safety and efficacy of nasal carbon dioxide for the treatment of pain and other symptoms related to temporomandibular disorders (TMD). Approximately 115 men and women ages 18 to 70 years old who have a history consistent with TMD-related pain for at least 3 months and meet all other eligibility criteria will be enrolled in this study. There may be up to two (2) visits to the clinic, screening and treatment. Screening and treatment may occur on the same day.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a history consistent with TMD-related pain for at least 3 months prior to screening
* Agree not to use certain medications prior to randomization within the study specified
* Females of childbearing potential must commit to using an acceptable method of birth control and have a negative pregnancy test.

Key Exclusion Criteria:

* Have recent history of alcohol or drug abuse within 2 years prior to randomization
* Current major psychiatric disorder such as suicidal ideation, bipolar, panic disorder, schizophrenic, or psychoses
* History of asthma (other than mild or intermittent)
* Have an existing serious unstable systemic disease (such as severe emphysema, other respiratory diseases, heart disease, etc.) that precludes participation in the study
* Clinically significant nasal disorder (such as deviated septum, presence of polyps, evidence of significant congestion, rhinitis, or other nasal abnormalities)
* Current diagnosis of fibromyalgia
* History or clear clinical evidence of osteoarthritis of temporomandibular joint (TMJ)
* A TMD diagnosis of disc displacement without reduction, "locking"

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in pain status from baseline over a 3 hour period | within 3 hours of the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Edward L. Truelove, DDS, MSD, Principal Investigator — University of Washington School of Dentistry
Locations (1):
- University of Washington, Department of Oral Medicine, Box 356370, Health Sciences Building, Seattle, Washington, United States